CLINICAL TRIAL: NCT04512053
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind Study of TAS-303 in Female Patients With Stress Urinary Incontinence
Brief Title: A Phase 2 Study of TAS-303 in Female Patients With Stress Urinary Incontinence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 10060070
Record Dates: First submitted 2020-08-07; First posted 2020-08-13 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Urinary Incontinence; Urinary Incontinence, Stress; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence; Lower Urinary Tract Symptoms | interventions — TAS-303

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAS-303 (Experimental)
  Interventions: Drug: TAS-303 18 mg/day
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TAS-303 18 mg/day — Oral administration for 12 weeks, once daily
  Arms: TAS-303
Drug: Placebo — Oral administration for 12 weeks, once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of TAS-303 in female patients with stress urinary incontinence.

DETAILED DESCRIPTION:
The main purpose of this study is to assess the efficacy of TAS-303 in female patients with stress urinary incontinence (SUI) compared with placebo as measured by the percent change in the average SUI episode frequency per 24 hours from baseline at week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient has symptoms of Stress Urinary Incontinence (SUI) for at least 12 weeks prior to study entry
* Urinary incontinence in the 1-hour pad weight test exceeds 2.0 g
* The average number of SUI episodes is 1 or more per day
* The average number of urge urinary incontinence (UUI) episodes is 0.43 or less per day
* The number of "SUI episodes" exceeds the number of "other episodes"
* The average number of urinary diurnal frequency is 10 or less per day and the average number of nocturia frequency is 2 or less per day

Key Exclusion Criteria:

* Patient has been diagnosed with mixed urinary incontinence (MUI) that is predominantly UUI
* Patient has treated medication or therapy for SUI within 14 days before prior to study entry
* Patient is considered to have SUI that would not be expected to improve unless treated with surgical therapy
* Patient had a history of surgical treatment for urinary incontinence (Trans-obturator tape surgery, Tension-free vaginal tape surgery, etc.)
* Patient has stage II or more of Pelvic Organ Prolapse (POP), or had a history of POP repair surgery within 180 days before prior to study entry
* Patient has a serious illness or medical condition

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
The percent change in the average SUI episode frequency per 24 hours | Baseline, week 12

SECONDARY OUTCOMES:
The average urinary incontinence episode frequency per 24 hours | Baseline, week 4, week 8, week 12
The urinary incontinence volume measured in a 24-hour pad test | Baseline, week 12
The change in the international Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) | Baseline, week 4, week 8, week 12
The change in the Patient's Global Impressions of Improvement (PGI I) questionnaire. | Baseline, week 4, week 8, week 12
The change in the incontinence quality of life instrument (I QOL) scores | Baseline, week 4, week 8, week 12
  The minimum score is 22 points and the maximum is 110 points. The higher scores mean a worse outcome.
The changes in the overactive bladder symptom score (OABSS) | Baseline, week 4, week 8, week 12
  The minimum score is 0 points and the maximum is 15 points. The higher scores mean a worse outcome.
Incidence of adverse events and side effects | Up to 13 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (4):
- Japan (4):
  - A site selected by Taiho Pharmaceutical Co., Ltd., Aichi
  - A site selected by Taiho Pharmaceutical Co., Ltd., Fukuoka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Osaka
  - A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Taiho Group (Taiho) provides a platform for accepting researchers requests for sharing anonymized, patient-level, analyzable datasets from articles published in peer-reviewed journals about the primary results from Taiho-sponsored interventional clinical trials in patients in which the medicine and the indication has received marketing approval from regulatory authorities in the United States, the European Union, and/or Japan on or after January 15, 2018.
  Access to the clinical trial data is contingent upon approval of a proposed study protocol by an independent review panel and the execution of a data-sharing agreement with the researcher.
  See: https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Takahashi S, Kato K, Yokoyama O, Takei M, Gotoh M. Efficacy and Safety of TAS-303 in Female Patients With Stress Urinary Incontinence: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Trial. J Urol. 2024 Aug;212(2):267-279. doi: 10.1097/JU.0000000000004024. Epub 2024 Jul 9. PMID 38979756